CLINICAL TRIAL: NCT01392677
Title: A 24-week, Multicentre, Randomised, Double-Blind, Placebo-Controlled, International Phase III Study With a 28-week Extension Period to Evaluate the Safety and Efficacy of Dapagliflozin 10mg Once Daily in Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control on a Background Combination of Metformin and Sulfonylurea
Brief Title: Evaluation of Safety and Efficacy of Dapagliflozin in Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Background Combination of Metformin and Sulfonylurea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1693C00005
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2013-12-27 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Mellitus; High HbA1c Level; Inadequate Glycaemic Control
Keywords: dapagliflozin; diabetes; hyperglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin 10 mg tablet (Experimental)
  Interventions: Drug: dapagliflozin
- matching placebo tablet (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dapagliflozin — 10 mg tablet, oral, once daily, 24- week treatment and 28- week extension period
  Arms: Dapagliflozin 10 mg tablet
Drug: placebo — matching placebo tablet, oral, once daily, 24- week treatment and 28- week extension period
  Arms: matching placebo tablet

SUMMARY:
This study intends to compare the efficacy and safety of dapagliflozin versus placebo in patients with type 2 diabetes who have inadequate glycaemic control on a background combination of metformin and sulfonylurea.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Men or women age ≥ 18 years old
* Stable dose combination of metformin and sulfonylurea
* HbA1c ≥7.7% and ≤11.0%

Exclusion Criteria:

* Type 1 diabetes mellitus or diabetes insipidus
* Recent cardiovascular events
* Kidney or urological disorders
* Hepatic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Johnsson, PhD, Medical Science Director, Study Director — AstraZeneca R&D, Global Medicines Development CVGI, SE-431 83 Mölndal, Sweden; Stephan Matthaei, Prof.Dr.med, Principal Investigator — Diabetes-Zentrum Quakenbruck
Locations (42):
- Canada (12):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney Mines, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Kensington, Prince Edward Island
  - Research Site, Laval, Quebec
  - Research Site, Québec, Quebec
- Czechia (6):
  - Research Site, Beroun
  - Research Site, České Budějovice
  - Research Site, Jílové u Prahy
  - Research Site, Prague
  - Research Site, Semily
  - Research Site, Vyškov
- Germany (6):
  - Research Site, Aßlar
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Falkensee
  - Research Site, Neuwied
  - Research Site, Pirna
- Poland (6):
  - Research Site, Kielce
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Zgierz
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Košice
  - Research Site, Považská Bystrica
  - Research Site, Rimavská Sobota
- Spain (8):
  - Research Site, Barcelona, Catalonia
  - Research Site, Santa Coloma de Gramanet (bcn), Catalu?a
  - Research Site, A Coruña, Galicia
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Oviedo
  - Research Site, Santa Coloma de Gramenet (bcn)

REFERENCES:
- [Derived] Matthaei S, Bowering K, Rohwedder K, Grohl A, Parikh S; Study 05 Group. Dapagliflozin improves glycemic control and reduces body weight as add-on therapy to metformin plus sulfonylurea: a 24-week randomized, double-blind clinical trial. Diabetes Care. 2015 Mar;38(3):365-72. doi: 10.2337/dc14-0666. Epub 2015 Jan 15. PMID 25592197
- See also: D1693C00005.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1200&filename=D1693C00005.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 24 Oct 2011. Last participant completed 24 week period: 07 Jan 2013. 311 participants were enrolled, 219 were randomized in 45 centers in 5 European countries and in North America. Men and women aged >= 18 years with inadequate glycemic control (HbA1c 7.0% to 10.5% prior to randomization).
Pre-assignment Details: During enrollment, diet and life-style advice was given to participants and was reinforced during a placebo lead-in period. Dose of anti-hyperglycemic combination therapy of metformin >= 1500 mg/day and maximum tolerated dose which must be at least half the maximum dose of sulfonylurea for at least 8 weeks prior to enrollment were to remain stable.
Groups:
- Placebo Plus Metformin Plus Sulfonylurea: Placebo once daily plus background combination of metformin and sulfonylurea
- Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea: Dapagliflozin 10mg once daily plus background combination of metformin and sulfonylurea
Period: Overall Study
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Started | 109 | 109
Completed | 101 | 101
Not Completed | 8 | 8
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Incorrect enrollment | 2 | 3
Not completed — Other reason | 3 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of study medication during the 24-week short-term double blind treatment period who have a non-missing baseline value and at least one post-baseline value for at least one efficacy variable to be analyzed at week 24.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea | Total
Number analyzed (Participants) | 108 | 108 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (9.24) | 61.1 (9.65) | 61.0 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 62 | 110
  Male | 60 | 46 | 106
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 102 | 104 | 206
  Black/African American | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Other | 1 | 1 | 2
Body Weight [Mean (Standard Deviation); unit: kg] | 90.07 (16.175) | 88.57 (17.584) | 89.32 (16.872)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.02 (4.581) | 31.93 (4.840) | 31.97 (4.702)
Glycosylated hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.24 (0.865) | 8.08 (0.912) | 8.16 (0.890)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 180.2 (43.13) | 167.4 (43.32) | 173.8 (43.61)
Fasting C-Peptide [Mean (Standard Deviation); unit: ng/mL] | 2.5 (0.98) | 2.5 (1.06) | 2.5 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in HbA1c Levels
Description: To compare the change from baseline in HbA1c to week 24 between dapagliflozin 10 mg in combination with metformin and sulfonylurea and placebo in combination with metformin and sulfonylurea.
Time Frame: Baseline to week 24
Population: Full Analysis Set, participants with non-missing baseline and week 24 values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Number analyzed (Participants) | 108 | 108
Percent | -0.17 [-0.31 to -0.02] | -0.86 [-1.00 to -0.72]
Statistical Analysis 1: Comparison: Placebo Plus Metformin Plus Sulfonylurea vs Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Significant at alpha=0.05 (2-sided). A hierarchical closed testing procedure was used to control Type I error across the primary & key secondary objectives; Longitudinal repeated measures model using mixed model with treatment group, baseline value, week and week*treatment and week*baseline; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.89 to -0.49], Standard Error of Mean 0.1022

2. Secondary Outcome: Adjusted Mean Change From Baseline in FPG
Description: To compare the change from baseline in fasting plasma glucose (FPG) to week 24 (LOCF) between dapagliflozin and placebo
Time Frame: Baseline to week 24
Population: Full Analysis Set, participants with non-missing baseline and week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Number analyzed (Participants) | 107 | 108
mg/dL | -0.78 [-7.56 to 6.01] | -34.23 [-40.98 to -27.48]
Statistical Analysis 1: Comparison: Placebo Plus Metformin Plus Sulfonylurea vs Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group as effect and baseline value as covariate; Mean Difference (Final Values) = -33.45, 95% CI 2-sided [-43.08 to -23.82], Standard Error of Mean 4.8846

3. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight
Description: To compare the change from baseline in total body weight to week 24 (LOCF) between dapagliflozin and placebo
Time Frame: Baseline to week 24
Population: Full Analysis Set, participants with non-missing baseline and week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Number analyzed (Participants) | 108 | 108
kg | -0.58 [-1.09 to -0.07] | -2.65 [-3.16 to -2.14]
Statistical Analysis 1: Comparison: Placebo Plus Metformin Plus Sulfonylurea vs Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group as effect and baseline value as covariate; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-2.79 to -1.35], Standard Error of Mean 0.3651

4. Secondary Outcome: Proportion of Participants With HbA1c Value < 7.0% at Week 24 (LOCF)
Description: To compare the proportion of subjects achieving a therapeutic glycemic response, defined as HbA1c <7.0%, at week 24 (LOCF) between dapagliflozin and placebo
Time Frame: Baseline to week 24
Population: Full Analysis Set, participants with non-missing baseline and week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Number analyzed (Participants) | 108 | 108
Percentage of participants | 11.1 [5.4 to 16.8] | 31.8 [23.3 to 40.2]
Statistical Analysis 1: Comparison: Placebo Plus Metformin Plus Sulfonylurea vs Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea; H0: proportion(treat) minus proportion (placebo) = 0 versus the alternative HA: proportion (treat) minus proportion (placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Based on methodology of Zhang, Tsiatis & Davidian and Tsiatis, Davidian, Zhang & Lu, with adjustment for baseline value; Risk Difference (RD) = 20.7, 95% CI 2-sided [10.7 to 30.6], Standard Error of Mean 5.056

5. Secondary Outcome: Adjusted Mean Change From Baseline in Seated Systolic Blood Pressure
Description: To compare the change from baseline in seated systolic blood pressure (SBP) to week 8 (LOCF) between dapagliflozin and placebo
Time Frame: Baseline to week 8
Population: Full Analysis Set, participants with non-missing baseline and week 8 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Number analyzed (Participants) | 105 | 105
mmHg | -0.27 [-2.60 to 2.05] | -4.04 [-6.36 to -1.72]
Statistical Analysis 1: Comparison: Placebo Plus Metformin Plus Sulfonylurea vs Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.025, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group as effect and baseline value as covariate; Mean Difference (Final Values) = -3.76, 95% CI 2-sided [-7.05 to -0.48], Standard Error of Mean 1.6677

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment plus 4/30 days or up to follow-up visit if earlier, or up to and including the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Placebo Plus Metformin Plus Sulfonylurea | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea
Serious Adverse Events (participants affected / at risk) | 6/109 | 1/109
Other Adverse Events (participants affected / at risk) | 7/109 | 5/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Metformin Plus Sulfonylurea (N=109) | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea (N=109)
aortic valve stenosis (Cardiac disorders) | 1 | 0
arrhythmia (Cardiac disorders) | 1 | 0
diabetic gangrene (Infections and infestations) | 1 | 0
sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
calculus ureteric (Renal and urinary disorders) | 1 | 0
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Metformin Plus Sulfonylurea (N=109) | Dapagliflozin 10mg Plus Metformin Plus Sulfonylurea (N=109)
urinary tract infection (Infections and infestations) | 7 | 5

LIMITATIONS AND CAVEATS:
For participants who did not complete 8 and/or 24 weeks, respectively, last observation carried forward (LOCF) was used for analyses of secondary endpoints. All endpoints were evaluated by excluding data after rescue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.